CLINICAL TRIAL: NCT05201261
Title: the Relationship Between Vertebral Body Length, Subarachnoid Space Width and Block Level
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Other Study IDs: block level
Record Dates: First submitted 2021-12-16; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-12

CONDITIONS: Combined Spinal Epidurai Anesthesia; Lower Extremity Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ultrasound-guided group: Adult patients with American Society of Anesthesiologists physical status I/II/III scheduled to undergo elective Lower limb surgery under spinal anesthesia were considered for eligibility.
  Interventions: Device: ltrasonic measure

INTERVENTIONS:
Device: ltrasonic measure — In the right decubitus position, the spine was scanned with an ultrasonic convex array probe. Starting from the sacrum, the length of each vertebral body of the lumbar spine was measured on a para-midsagittal oblique view. The intervertebral space was located and the width of the subarachnoid space was measured on a midsagittal and transverse view.

SUMMARY:
Spinal anesthesia technology has been widely used in various surgeries and multi-mode analgesia. Spinal ultrasound imaging has been proved to be a reliable tool for evaluating spinal parameters. Ultrasound-guided spinal puncture technology has also been skillfully applied in clinical practice. How to provide perfect nerve block effect for operation, provide good postoperative analgesia, and prevent unnecessary extensive block leading to other complications and related risks has always been the focus of anesthesiologists. Doses and the relationship between the anesthesia plane great individual differences, and previous research on the patient's own condition such as height, weight, 6 to the anesthesia plane have different results, the influence of clinical work often refer patients height adjustment of drug doses, this research attempts to evaluate ultrasound was used to assess spinal vertebral body in the plane of the length and width of subarachnoid and anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective lower limbs surgery
* ASA: grade I to III

Exclusion Criteria:

* There are contraindications to spinal anesthesia
* Allergic to local anesthetics
* Patient refused

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective surgery under spinal anesthesia. Inclusion criteria: (1) Elective lower extremity surgery; (3) ASA (American Society of Anesthesiologists) Grading: ⅰ - ⅲ.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
The length of lumbar cone | 1year
  Ultrasound findings
The width of subarachnoid space was measured by ultrasound | 1year
  Ultrasound findings